CLINICAL TRIAL: NCT06268626
Title: Minimally Invasive Strategies for Early Detection of Uterine Cancer in Patients With Abnormal Uterine Bleeding
Brief Title: Detection of Endometrial Cancer Through Risk Modelling
Acronym: DETECTR
Status: Not yet recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Aline Talhouk, Principal Investigator, University of British Columbia
Other Study IDs: H22-02426; F22-01302 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR)); F21-03695 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2024-01-30; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Endometrial Cancer
Keywords: Screening; Prevention; Women's Health; Reproductive health; Abnormal Uterine Bleeding
MeSH Terms: conditions — Endometrial Neoplasms; Metrorrhagia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal DNA Vaginal microbiome Vaginal pH Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- EIN/EC BIOPSY RESULT: Vaginal DNA, microbiome, pH, and saliva samples sequenced. Participation ends here.
- EH BIOPSY RESULT: Vaginal DNA, microbiome, pH, and saliva samples sequenced. All invited to move on to Part B and samples sequenced for 6 additional months.
- NEGATIVE BIOPSY RESULT: Control for natural and spontaneous changes in vaginal DNA, microbiome, pH, and saliva samples sequenced.
  Random subset selected to move on to Part B and samples sequenced for 6 additional months.

SUMMARY:
The goal of this study is to combine information on risk factors from health questionnaires with minimally invasive biological tests (vaginal DNA and microbiome swabs, pH, hormones) to predict the risk of endometrial cancer (EC), better understand progression of the disease, and identify opportunities for intervention.

This study will recruit patients who are already scheduled to undergo diagnostic evaluation for abnormal uterine bleeding via endometrial biopsy. In Part A, consented participants will be asked to fill out an online risk factor questionnaire. Samples will be collected by the gynecologist at the biopsy appointment. After biopsy results are obtained, all samples from participants diagnosed with EC or precursors, plus a random subset with benign results, will be selected to be sequenced and analyzed.

In Part B, that subset of selected non-malignant participants, based on biopsy, will be invited to take part in lifestyle tracking using a Fitbit, questionnaires, and to provide another round of at-home vaginal samples to identify any persistent genetic mutations or microbiome alterations 6-8 months later.

DETAILED DESCRIPTION:
Study Part A

1. Gynecologist Visit

   1. Patients over the age of 40 who are scheduled for an appointment for diagnostic evaluation of abnormal uterine bleeding (AUB) with one of the gynecologist study partners, will be invited to participate in this study. Those who consent to participate and undergo a uterine biopsy, which is the standard of care for AUB, will be enrolled in the study.
   2. If a biopsy was not anticipated when the appointment was scheduled and therefore the patient was unable to provide consent prior to their appointment, the gynecologist will explain the study and obtain verbal consent to collect the samples and provide the patient's contact information to the study coordinator. The coordinator will contact the patient as soon as possible to explain the study and obtain informed consent.
2. Primary Sample Collection

   1. During the standard biopsy procedure, the gynecologist will also collect study specific samples including: swabs for vaginal DNA and microbiome samples, a pH litmus test strip, and a saliva sample kit.
   2. Participants will consent to have their electronic medical records including biopsy results shared with the study team as part of the study. A member of the study team will further call the location where the endometrial biopsy occurred to ask for any remaining specimen that could be used for comparison to the vaginal swab DNA sequencing, as indicated on the consent form.
3. Email - REDCap Risk Questionnaire

   a. Participants will receive an email from a study coordinator with a link to a REDCap epidemiological risk questionnaire. The 5-10 minute survey will provide the information needed to compute their absolute risk of being diagnosed with EC in the next 5 years. Absolute risks will be calculated using the validated Pfeiffer et al. model (PMID 23935463).

   Study Part B
4. Selection, Consent and MyCap Enrolment

   1. After the biopsy results are reviewed, participants will be selected to have their specimen from Part A sequenced and analyzed. For budget reasons, only those participants diagnosed with endometrial cancer or hyperplasia (with or without atypia) will be sequenced and analyzed, along with twice as many randomly selected participants with benign diagnoses.
   2. Participants diagnosed with EC or endometrial intraepithelial neoplasia (EIN) will likely be recommended a hysterectomy, as per standard of care, and will be ineligible to continue in the next phase, since they will no longer be at risk for uterine cancer.
   3. All remaining participants diagnosed with endometrial hyperplasia (EH) without atypia and the non-malignant biopsy participants who were selected for sequencing will be contacted to participate in Study Part B. The study coordinator will explain this portion of the study and the procedures involved. If the participant is interested, the study coordinator will assist them in downloading MyCap, a mobile app integration for REDCap to register for the study and provide electronic consent. Participants will be mailed a Fitbit fitness tracker to monitor their lifestyle, activity and sleep patterns, along with instructions on how to set it up. They will be asked to manually report daily step counts and sleep data from their FitBit into MyCap app until the time of their second sample collection, at least 6 months later.
5. Second Sample Collection

   1. After approximately 6-8 months, participants will receive an at-home collection kit in the mail with a tampon and swab for DNA collection along with a vaginal microbiome sampling kit, a vaginal pH testing kit, and a saliva kit (n~200). The investigators will ask that participants not have sexual intercourse, use vaginal medications, feminine sprays, douches, genital wipes or contraceptive spermicides for at least 48 hours before providing sample collection.

      * Tampon and swab #1: DNA will be collected from a tampon worn for 6-8 hours as well as by self-sample using a vaginal swab.
      * Swab #2: Vaginal microbiome samples will be obtained with a second vaginal swab using the DNAGenotek Inc. OMNIgene vaginal collection kit.
      * pH measurement: The pH kit will contain an indicator strip and a reference colour sheet; participants will be asked to take a photo of the strip next to the reference colour sheet as well as record the result in MyCap.
      * Saliva: A saliva collection kit (Affinity Diagnostics) will be used for hormone measurements and additional DNA extraction, if necessary.
   2. Participants will be provided with a postage paid return mailing envelope to send the samples. They will be prompted through MyCap to indicate when they receive their kits, when they are completed, and when they are mailed back.
6. Molecular Analysis and Results

   1. All samples will be processed and stored for follow-up investigations by batch. The investigators will prioritize genetic sequencing and screening of samples from participants in which the investigators observed cancer-associated DNA mutations in samples collected in Part A.
   2. It is important to understand that genetic mutations or alterations are fairly common in patients with abnormal uterine bleeding; and the majority will resolve on their own after shedding of the uterine lining. Because of this, and the fact that these initial analyses are experimental and are done for research purposes only, genetic results will not be communicated to participants. The significance of genetic mutations or microbiome alterations is not yet interpretable at this stage in the investigator's research.
   3. However, if the investigators discover that the same specific mutations or microbiome alterations are persistent in the second vaginal samples collected 6-8 months later, the participant and their gynecologist will be notified. The treating gynecologist will determine what, if any, follow-up or monitoring is appropriate.

8) Exit Survey

a. Participants, depending on the stage at which they exit the study, will be asked about their experience with the sample collection during biopsy, the risk questionnaire, the MyCap app, and the at-home sample collection.

ELIGIBILITY:
Inclusion Criteria:

Study Part A:

* 40 years and older
* Experiencing unexplained abnormal uterine bleeding (i.e., not from IUD, etc.)
* Have an intact uterus
* Referred for an endometrial biopsy

Study Part B:

* Those selected for sequencing (from Part A) and who retained their uterus.

Exclusion Criteria:

Study Part A:

* Endometrial sampling, pelvic radiation, or vaginal infection (vaginosis, yeast) in the past 3 months
* Started hormone therapy (HRT, birth control, IUD) in the past year (with the exception of tamoxifen)
* Intercourse, vaginal product use, or douching in the past 48 hours

Study Part B:

* Same as Study Part A
* EC or EIN, or anyone who is recommended a hysterectomy

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study investigators will have 10-15 study gynecologists across British Columbia, Canada, who will be recruiting study participants from patients who are referred to them for an endometrial biopsy due to abnormal uterine bleeding. The investigators aim to recruit ~1000 participants in Study Part A in order to achieve their target sample size of n=50 EIN/EC and n=150 EH.
  Sequenced participants will be invited to participant in Study Part B and provide additional samples.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Association Between Risk Factor Data and Endometrial Cancer and It's Precursors. | Through study completion, anticipated 1-2 years
  Participants will receive an email from a study coordinator with a link to a REDCap epidemiological risk questionnaire. The 5-minute survey will provide the information needed for the investigators to compute and assign each participant an absolute risk score of being diagnosed with endometrial cancer in the next 5 years from the time of data collection. Absolute risks will be calculated using the validated Pfeiffer et al. model, which has been externally validated.
Change in Risk Prediction of Endometrial Cancer When Mutation and Microbiome Data Is Combined With Traditional Risk Factors, Compared to Traditional Risk Factors Alone. | Through study completion, anticipated 1-2 years
  At the time of the endometrial biopsy procedure, the study gynecologist will collect vaginal DNA using a swab, vaginal microbiome using a swab, vaginal pH using a litmus kit, and saliva for hormone analysis. Vaginal microbiome samples and pH will be collected using the DNAGenotek OMNIgene vaginal kit and GYNEX pHem-Alert vaginal kits. Saliva will be collected using saliva kit (Affinity Diagnostics).
  Participants will consent to have their electronic medical records including biopsy results shared with the study team as part of the study. A member of the study team will further call the location where the endometrial biopsy occurred to ask for any remaining specimens that could be used for comparison to the vaginal swab DNA sequencing, as indicated on the consent form.
  Epidemiological risk factors will be integrated with mutations and microbiome signatures from uterine/vaginal sampling to predict the presence of endometrial cancer and its precursors.
Persistence of Mutations and Microbiome Alterations in Participants With Endometrial Hyperplasia. | Through study completion, anticipated 1-2 years
  Participants will be asked to self-collect vaginal specimens for DNA and microbiome analysis, test vaginal pH using an at-home collection kit, and obtain a saliva sample. For DNA collection, participants will be asked to self-sample using a vaginal swab as well as wear a tampon for 6-8 hours. For the vaginal microbiome sampling, participants will obtain a second self-sampled vaginal swab using the DNAGenotek Inc. OMNIgene vaginal collection kit. The pH kit will contain an indicator strip and a reference colour sheet. Participants will be asked to complete a saliva kit (Affinity Diagnostics).
  Approximately 6 months later, participants will be asked to repeat self-collection.
  Self-collected participant data will be utilized to assess the proportion of persistent endometrial cancer-associated mutations in those with endometrial hyperplasia compared to other non-malignant conditions in females with abnormal uterine bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Aline Talhouk, PhD, Principal Investigator — University of British Columbia; Anna Tinker, MD, Principal Investigator — University of British Columbia
Locations (1):
- VGH Research Pavilion, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pfeiffer RM, Park Y, Kreimer AR, Lacey JV Jr, Pee D, Greenlee RT, Buys SS, Hollenbeck A, Rosner B, Gail MH, Hartge P. Risk prediction for breast, endometrial, and ovarian cancer in white women aged 50 y or older: derivation and validation from population-based cohort studies. PLoS Med. 2013;10(7):e1001492. doi: 10.1371/journal.pmed.1001492. Epub 2013 Jul 30. PMID 23935463